CLINICAL TRIAL: NCT05474820
Title: Saliva Irisin Level is Higher and Related With Interleukin 6 in Generalized Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Nur Balci, DDs, PhD, ASSOC. PROF DR, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 361
Record Dates: First submitted 2022-07-23; First posted 2022-07-26 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-07

CONDITIONS: Inflammatory Response; Periodontitis
Keywords: periodontitis; irisin
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saliva and serum collection of patients and samples molecules analysis (Other): After periodontal examination, samples were collected from all patients via informing them about procedures. Then all samples were stored at -80 C unto analyses.
  Interventions: Other: Samples collection and ELISA analyses; Diagnostic Test: Evaluating periodontal paramètres
- Periodontal examination (Other): All periodontal indices were measured in six sites in each tooth present in the arch by one calibrated periodontist
  Interventions: Other: Samples collection and ELISA analyses; Diagnostic Test: Evaluating periodontal paramètres

INTERVENTIONS:
Other: Samples collection and ELISA analyses — The serum and unstimulated saliva samples were taken from all patients between 8:00 and 10:00 in the morning. Saliva samples were centrifuged at 10,000 rpm (10 min) whereas venous blood samples were centrifuged at 4000 rpm for 10 min.
  For the analysis of irisin and IL-6 specific ELISA Kits (Elabscience, Houston, Texas, USA) were used to determine the molecules in both serum and saliva samples in accordance with the manufacturer's instructions. All samples were run in duplicate, and values have been averaged.
Diagnostic Test: Evaluating periodontal paramètres — The clinical periodontal parameters (plaque index (PI), probing pocket depth (PD), gingival recession (GR), clinical attachment loss (CAL), and bleeding on probing (BOP)) were recorded on periodontal charts in each patient

SUMMARY:
Irisin is novel adipomyokine known as a mediator of physical activity that produced mainly by skeletal muscle and adipose tissues. It is cleaved from the fibronectin type III domain-containing protein 5 (FDNC5), which is, in turn, induced by peroxisome proliferator-activated receptor-ɣ co-activator 1-α (PGC-1α). Several studies reported that irisin is related with pathogenesis of many diseases which are known to be associated with periodontal disease such as obesity, diabetes mellitus, rheumatoid arthritis, cardiovascular disease, nonalcoholic fatty liver disease and metabolic bone diseases. There are several studies those have reported that increased IL-6 levels are associated with progression and severity of periodontitis . Recently, it has been shown that irisin is expressed in human periodontal ligament cells (hPDL), dental pulp stem cells and osteoblasts. Also, a few studies revealed that irisin promotes growth, migration and matrix formation in hPDL cells and cementoblast differentiation. To the best our knowledge, there 's one study has been reported that the higher levels of irisin in saliva in patient with chronic periodontitis

DETAILED DESCRIPTION:
Twenty systemically healthy subjects with healthy periodontium and 20 patients with stage III grade B generalized periodontitis were enrolled for this cross-sectional study. The study was performed in accordance with the Helsinki Declaration of 1975, as revised in 2013. Before starting, the informed consent was obtained from all participants which was approved by the human subject's ethics board of Istanbul Medipol University's Faculty of Dentistry for use and access of human subjects in research.For all study subjects, the exclusion criteria were (1) use of contraceptive drugs; (2) use of antibiotics, anti-inflammatory drugs, or immunosuppressants in the last 3 months before the study; (3) alcohol consumption; (4) pregnancy or breastfeeding; (5) taking drugs that could cause side effects such as gingival hypertrophy or hyperplasia; and (6) any periodontal treatments in the 3 months prior to enrollment. All participants were systemically healthy and non-smokers (never smokers).The clinical periodontal parameters (plaque index (PI), probing pocket depth (PD), gingival recession (GR), clinical attachment loss (CAL), and bleeding on probing (BOP)) were recorded on periodontal charts in each patient .For the analysis of irisin and IL-6 specific ELISA Kits (Elabscience, Houston, Texas, USA) were used to determine the molecules in both serum and saliva samples in accordance with the manufacturer's instructions. The minimum detectable doses of irisin and IL-6 for saliva with these assay kits were 1,28 and 13,22 pg/ml, respectively. For serum, minimum detectable irisin dose was 175,43 whereas IL-6 was 0,06 pg/ml. All samples were run in duplicate, and values have been averaged.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* clinical diagnosis of periodontitis
* clinical diagnosis of periodontal health

Exclusion Criteria:

*history of regular use of systemic antibiotics anti-inflammatory, or antioxidant drugs (previous 3 months)

* nonsurgical periodontal treatment (previous 6 months)
* surgical periodontal treatment (previous 12 months)
* presence of<10 teeth
* current medications affecting gingival health (calcium channel blockers, phenytoin, cyclosporine, and hormone replacement therapy)
* diabetes
* diagnosis of rheumatoid arthritis
* pregnancy
* lactating
* smoking
* excessive alcohol consumption.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Pocket probing depth | 3 months
  Measurement of the depth of a sulcus or periodontal pocket determined by measuring distance from a gingival margin to the base of the sulcus or pocket with a calibrated periodontal probe.
Clinical attachment level | 3 months
  Clinical attachment level (or loss, CAL) is a more accurate indicator of the periodontal support around a tooth than probing depth alone. CAL is measured from a fixed point on the tooth that does not change, the CEJ.
  To calculate CAL, two measurements are needed: distance from the gingival margin to the CEJ and probing depth.
  In recession: probing depth (+) gingival margin to the CEJ (add). In tissue overgrowth: probing depth (-) gingival margin to the CEJ (subtract)

SECONDARY OUTCOMES:
Saliva and serum samples processing and analyses | 1 month
  Saliva and serum samples obtained for each patient were used for cytokine analysis. Prepared samples were analyzed for Irisin and IL-6 via ELISA kits.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, School of Dentistry, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Pullisaar H, Colaianni G, Lian AM, Vandevska-Radunovic V, Grano M, Reseland JE. Irisin promotes growth, migration and matrix formation in human periodontal ligament cells. Arch Oral Biol. 2020 Mar;111:104635. doi: 10.1016/j.archoralbio.2019.104635. Epub 2019 Dec 16. PMID 31869727